CLINICAL TRIAL: NCT06257563
Title: Co-developing a Bio-experiential Approach and Intervention to Support the Mental Health and Well-being of Dementia Patients and Their Caregivers at Home (TEND)
Brief Title: Toolkit for Experiential Well-beiNg in Dementia (TEND)
Acronym: TEND
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are withdrawing our study due to regulatory requirements from our funding source.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Christine S. Ritchie, MD, MPH, Director of Research, Division of Palliative Care and Geriatric Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022P001401
Record Dates: First submitted 2024-01-19; First posted 2024-02-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Bio-Experiential; Videogame; Psychosocial
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: All dyads will use the "Isle of TEND" videogame platform for 20-30 minutes three-four times a week for four weeks. The Isle of TEND is supported on computers and laptops and is accessible through a link on any modern browser window.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isle of TEND Intervention (Experimental): All participants will engage in the Isle of TEND Intervention.
  Interventions: Other: Isle of TEND Intervention

INTERVENTIONS:
Other: Isle of TEND Intervention — The "Isle of TEND" is an interactive videogame platform in which users navigate to different modules on a virtual island. The modules aim to create a pleasant, shared and "error-free" experience for persons with dementia and their caregivers.

SUMMARY:
The goal of this project is to conduct an open pilot (N=5) among dyads (persons living with dementia and their caregivers) to assess the preliminary effects of an online videogame platform. The "Isle of TEND" is an immersive and interactive videogame platform designed for persons living with dementia and their caregivers. Dyads will use the platform three to four times a week for 20-30 minutes across four weeks. The investigators will assess for improvements in relationship satisfaction, wellbeing, and positive emotions and gather feedback on engagement in the platform. Dyads will complete measures at baseline and post-intervention as well as brief measures after each platform use.

DETAILED DESCRIPTION:
The aim of this phase is to assess initial active engagement, sustained attention, and positive emotions of the "Isle of TEND" intervention platform. Our participants (N = 5 dyads) will be persons living with moderate-severe dementia and their caregivers in the Boston area.

The intervention, "Isle of TEND" is an immersive and interactive videogame platform designed for persons living with dementia and their caregivers. Studio Elsewhere, a design and development team, developed the platform in consideration with feedback generated from focus groups and design workshops. Users navigate the online island and explore accompanying modules with varying audio and visual features. The platform aims to engage dyads in an enjoyable, shared, and "error-free" experience (i.e., creating poetry, viewing virtual art).

Participants will use their personal "travel journal" after each platform session, in which they log engagement and positive emotion. Dyads are also encouraged to provide free response feedback on the platform. Once a week, dyads will record themselves as they use the platform. The investigators will conclude the pilot with exit interviews. Baseline and post intervention assessments will include self-reported measures including relationship satisfaction, wellbeing, and caregiver stress. The research team will engage in behavioral observation coding to assess active engagement.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver (specifically, a family member) of a person with moderate-severe dementia and person with moderate-severe dementia
* Moderate to severe as determined by Functional Assessment Staging Tool (FAST Scale) taken by caregiver
* Age 18 or older
* English-speaking
* Willing and able to use the platform together 3-4 times a week for 20-30 minutes
* Located in the Boston area

Exclusion Criteria:

* Lack of access to internet and/or a computer with a camera
* Untreated serious mental illness and or substance use diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Engagement | 4 weeks
  The investigators will examine whether the Isle of TEND is able to capture engagement among participants. Participants will complete the User Engagement Scale after each platform use to report engagement.
  The User Engagement Scale is on a scale of 1 (Strongly disagree) to 5 (Strongly agree) with higher scores indicating greater engagement. Participants can score between 3 and 15.
Adherence | 4 weeks
  The investigators will measure adherence through objective and self report measures. Participants will log in a journal each time and duration they use the platform. Additionally, the website platform will run diagnostics to report aggregated use across all participants.

SECONDARY OUTCOMES:
Depression | 4 weeks
  The investigators will measure depression through the Geriatric Depression Scale. Participants will complete the Geriatric Depression Scale at baseline and post test periods.
  The Geriatric Depression Scale (GRS) is on a Yes/No scale. A score greater than 5 indicates depression. Participants can score between 0 and 15.
Caregiver stress | 4 weeks
  The investigators will examine measure caregiver stress through the Modified Caregiver Stress Index. Participants will complete the MCSI at baseline and post test periods.
  The Modified Caregiver Stress Index (MCSI) is on a scale of 2 (Yes, on a Regular Basis) to 0 (No). A higher score indicates greater caregiver stress. Participants can score between 0 and 26.
Relationship Satisfaction | 4 weeks
  The investigators will examine measure relationship satisfaction through the Dyadic Relationship Scale. Participants will complete the DRS at baseline and post test periods.
  The Dyadic Relationship Scale (DRS) is on a scale of 0 (Strongly Agree) to 3 (Strongly Disagree). A higher score indicates greater relationship satisfaction. Participants can score between 0 and 33.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ritchie, MD, MSPH, Principal Investigator — Massachusetts General Hospital; Ana-Maria Vranceanu, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rochon EA, Sy M, Phillips M, Anderson E, Plys E, Ritchie C, Vranceanu AM. Bio-Experiential Technology to Support Persons With Dementia and Care Partners at Home (TEND): Protocol for an Intervention Development Study. JMIR Res Protoc. 2023 Dec 29;12:e52799. doi: 10.2196/52799. PMID 38157239
- [Background] Gitlin LN, Winter L, Dennis MP, Hodgson N, Hauck WW. A biobehavioral home-based intervention and the well-being of patients with dementia and their caregivers: the COPE randomized trial. JAMA. 2010 Sep 1;304(9):983-91. doi: 10.1001/jama.2010.1253. PMID 20810376
- [Background] Poon E. A Systematic Review and Meta-Analysis of Dyadic Psychological Interventions for BPSD, Quality of Life and/or Caregiver Burden in Dementia or MCI. Clin Gerontol. 2022 Jul-Sep;45(4):777-797. doi: 10.1080/07317115.2019.1694117. Epub 2019 Nov 22. PMID 31752633
- [Background] Sorensen S, Duberstein P, Gill D, Pinquart M. Dementia care: mental health effects, intervention strategies, and clinical implications. Lancet Neurol. 2006 Nov;5(11):961-73. doi: 10.1016/S1474-4422(06)70599-3. PMID 17052663
- [Background] Gilhooly KJ, Gilhooly ML, Sullivan MP, McIntyre A, Wilson L, Harding E, Woodbridge R, Crutch S. A meta-review of stress, coping and interventions in dementia and dementia caregiving. BMC Geriatr. 2016 May 18;16:106. doi: 10.1186/s12877-016-0280-8. PMID 27193287
- [Background] Cheng Z, Zhou M, Sabran K. Mobile app-based interventions to improve the well-being of people with dementia: a systematic literature review. Assist Technol. 2024 Jan 2;36(1):64-74. doi: 10.1080/10400435.2023.2206439. Epub 2023 May 11. PMID 37115814
- [Background] Cardona JS, Lopez JA, Vela FLG, Moreira F. Meaningful learning: motivations of older adults in serious games. Univers Access Inf Soc. 2023 Mar 14:1-16. doi: 10.1007/s10209-023-00987-y. Online ahead of print. PMID 37361677
- [Background] Huang LC, Yang YH. The Long-term Effects of Immersive Virtual Reality Reminiscence in People With Dementia: Longitudinal Observational Study. JMIR Serious Games. 2022 Jul 25;10(3):e36720. doi: 10.2196/36720. PMID 35877169
- [Background] Astell AJ, Bouranis N, Hoey J, Lindauer A, Mihailidis A, Nugent C, Robillard JM; Technology and Dementia Professional Interest Area .... Technology and Dementia: The Future is Now. Dement Geriatr Cogn Disord. 2019;47(3):131-139. doi: 10.1159/000497800. Epub 2019 Jun 27. PMID 31247624